CLINICAL TRIAL: NCT02200211
Title: Study of Binocular Computer Activities for Treatment of Amblyopia
Acronym: ATS18
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Pediatric Eye Disease Investigator Group (Network); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATS18; 2U10EY011751 (NIH)
Record Dates: First submitted 2014-07-23; First posted 2014-07-25 (Estimated); Results first posted 2018-10-15 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Amblyopia
Keywords: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Binocular Treatment (Experimental): Binocular computer game play 1 hour per day, 7 days per week (minimum of 4 days per week)
  Interventions: Device: iPad®
- Patching Treatment (Active Comparator): Patching 2 hours per day, 7 days per week
  Interventions: Other: Patching 2 hours per day, 7 days per week

INTERVENTIONS:
Device: iPad® — Binocular therapy on iPad®
  Arms: Binocular Treatment
Other: Patching 2 hours per day, 7 days per week
  Other Names: Patching
  Arms: Patching Treatment

SUMMARY:
The purpose of the study is to compare the effectiveness of 1 hour/day of binocular game play 7 days per week with 2 hours/day patching 7 days per week in children 5 to <17

DETAILED DESCRIPTION:
The purpose of the study is to 1) compare the effectiveness of 1 hour/day of binocular game play 7 days per week (minimum of 4 days per week) with 2 hours/day patching 7 days per week, in children 5 to <13 years of age (younger cohort), as a non-inferiority study; and 2) to compare the effectiveness of 1 hour/day of binocular game play 7 days per week (minimum of 4 days per week) with 2 hours/day patching 7 days per week, in children 13 to <17 years of age (older cohort), as a superiority study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 5 to <17 years
2. Amblyopia associated with strabismus, anisometropia, or both (previously treated or untreated)

   1. Criteria for strabismus: At least one of the following must be met:

      * Presence of a heterotropia on examination at distance or near fixation (with or without spectacles)
      * Documented history of strabismus which is no longer present (which in the judgment of the investigator could have caused amblyopia)
   2. Criteria for anisometropia: At least one of the following criteria must be met:

      * ≥0.50 diopter (D) difference between eyes in spherical equivalent
      * ≥1.50 D difference between eyes in astigmatism in any meridian
   3. Criteria for combined-mechanism amblyopia: Both of the following criteria must be met:

      * Criteria for strabismus are met (see above)
      * ≥1.00 D difference between eyes in spherical equivalent OR ≥1.50 D difference between eyes in astigmatism in any meridian
      * Note: the spherical equivalent requirement differs from that in the definition for refractive/anisometropic amblyopia
3. No amblyopia treatment in the past 2 weeks (patching, atropine, Bangerter, vision therapy)
4. Refractive correction (spectacles or contact lenses, if applicable) must meet the following criteria at enrollment and be based on a cycloplegic refraction that is not more than 7 months old.

   1. Requirements for Correction of Refractive Error:

      1. For subjects meeting criteria for strabismic (only) amblyopia (see 2.2.1 #2 above):

         • Hypermetropia, if corrected, must not be under-corrected by more than +1.50 D spherical equivalent, and the reduction in plus sphere must be symmetric in the two eyes.
      2. For subjects meeting criteria for anisometropic or combined-mechanism amblyopia (see 2.2.1 #2 above):

         * Spherical equivalent must be within 0.50 D of fully correcting the anisometropia
         * Hypermetropia must not be under-corrected by more than +1.50 D spherical equivalent, and reduction in plus must be symmetric in the two eyes
         * Cylinder power in both eyes must be within 0.50 D of fully correcting the astigmatism
         * Cylinder axis for both eyes must be within 6 degrees of the axis of the cycloplegic refraction when cylinder power is ≥1.00 D
   2. Refractive corrections meeting the above criteria must be worn for either:

      * 16 weeks or more or
      * Until visual acuity in amblyopic eye is stable (defined as 2 consecutive visual acuity measurements by the same testing method at least 4 weeks apart with <1 line change (<5 letters if E-ETDRS))
   3. Monocular or binocular contact lens wear is allowed provided the contact lenses meet the above refractive requirements at the corneal plane. The same form of correction must be worn throughout the entire study during study procedures (i.e., no changing between contacts and spectacles while patching or while game-playing or study testing). Safety glasses are not required for subjects wearing contact lenses, but investigators are encouraged to suggest safety glasses be worn over contact lenses.
5. Visual acuity, measured in each eye without cycloplegia in current refractive correction (if applicable) within 7 days prior to randomization using the Amblyopia Treatment Study single-surround HOTV (ATS-HOTV) visual acuity protocol for children < 7 years and the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity protocol for children ≥ 7 years on a study-approved device displaying single surrounded optotypes, as follows:

   1. Visual acuity in the amblyopic eye 20/40 to 20/200 inclusive (33 to 72 letters if E-ETDRS)
   2. Visual acuity in the fellow eye 20/25 or better (≥ 78 letters if E-ETDRS)
   3. Interocular difference ≥ 3 logMAR lines (≥ 15 letters if E-ETDRS) (i.e., amblyopic-eye acuity at least 3 logMAR lines worse than fellow-eye acuity)
6. Heterotropia or heterophoria with a total near deviation of ≤ 10∆ (measured by PACT).
7. Ability to align the nonius cross on the binocular game system (angles of ocular deviation >10∆ would require the nonius cross to be adjusted to such an extent that playing of the game would be compromised).
8. Subject is able to play Hess Falling Blocks game on the study iPad® (on easy setting) under binocular conditions (with red-green glasses), as demonstrated by scoring at least 1 line in the office.
9. Investigator is willing to prescribe computer game play or patching per protocol.
10. Parent understands the protocol and is willing to accept randomization.
11. Parent has phone (or access to phone) and is willing to be contacted by Jaeb Center staff.
12. Relocation outside of area of an active Pediatric Eye Disease Investigator Group (PEDIG) site for this study within the next 16 weeks is not anticipated.

Exclusion Criteria:

A subject is excluded for any of the following reasons:

1. Prism in the refractive correction at time of enrollment (eligible only if prism is discontinued 2 weeks prior to enrollment).
2. Myopia greater than -6.00 D spherical equivalent in either eye.
3. Previous intraocular or refractive surgery.
4. Any treatment for amblyopia (patching, atropine, Bangerter filter, or vision therapy) during the past 2 weeks. Previous amblyopia therapy is allowed regardless of type, but must be discontinued at least 2 weeks immediately prior to enrollment.
5. Ocular co-morbidity that may reduce visual acuity determined by an ocular examination performed within the past 7 months (Note: nystagmus per se does not exclude the subject if the above visual acuity criteria are met).
6. No Down syndrome or cerebral palsy
7. No severe developmental delay that would interfere with treatment or evaluation (in the opinion of the investigator). Subjects with mild speech delay or reading and/or learning disabilities are not excluded.
8. Heterotropia or heterophoria with a total ocular deviation >10∆ (phoria plus tropia >10∆) at near (measured by PACT).

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 485 (Actual)
Dates: Start 2014-09-11 (Actual); Primary Completion 2016-08-19 (Actual); Study Completion 2016-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Holmes, MD, Study Chair — Mayo Clinic; Vivan Manh, OD, Study Chair — University of Washington
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Seattle Children's Hospital, University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH data sharing policy, a de-identified database is placed in the public domain on the PEDIG public website after the completion of each protocol and publication of the primary manuscript.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After primary manuscripts are published
Access Criteria: Users accessing the data must enter an email address.

REFERENCES:
- [Result] Holmes JM, Manh VM, Lazar EL, Beck RW, Birch EE, Kraker RT, Crouch ER, Erzurum SA, Khuddus N, Summers AI, Wallace DK; Pediatric Eye Disease Investigator Group. Effect of a Binocular iPad Game vs Part-time Patching in Children Aged 5 to 12 Years With Amblyopia: A Randomized Clinical Trial. JAMA Ophthalmol. 2016 Dec 1;134(12):1391-1400. doi: 10.1001/jamaophthalmol.2016.4262. PMID 27812703
- [Derived] Tailor V, Ludden S, Bossi M, Bunce C, Greenwood JA, Dahlmann-Noor A. Binocular versus standard occlusion or blurring treatment for unilateral amblyopia in children aged three to eight years. Cochrane Database Syst Rev. 2022 Feb 7;2(2):CD011347. doi: 10.1002/14651858.CD011347.pub3. PMID 35129211
- See also: PEDIG Public Website — http://www.pedig.net

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two separate sub-studies based on age at enrollment
  Younger Cohort defined as 5 to <13 years of age Older Cohort defined as 13 to <17 years of age
Groups:
- Binocular Treatment Younger; Binocular Treatment Older: Binocular computer game play 1 hour per day, 7 days per week (minimum of 4 days per week)
  iPad®: Binocular therapy on iPad®
- Patching Treatment Younger; Patching Treatment Older: Patching 2 hours per day, 7 days per week
Period: Overall Study
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger | Binocular Treatment Older | Patching Treatment Older
Started | 190 | 195 | 40 | 60
Included in 16-week Primary Analysis (16-week visits completed within pre-specified analysis window (148-196 days after randomization)) | 177 | 186 | 39 | 56
Completed (Completed 16-week study) | 182 | 188 | 39 | 58
Not Completed | 8 | 7 | 1 | 2
Not completed — Lost to Follow-up | 7 | 7 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Binocular Treatment Younger Cohort (5 to <13 Years); Binocular Treatment Older Cohort (13 to <17 Years): Binocular computer game play 1 hour per day, 7 days per week (minimum of 4 days per week)
  iPad®: Binocular therapy on iPad®
- Patching Treatment Younger Cohort (5 to <13 Years); Patching Treatment Older Cohort (13 to <17 Years): Patching 2 hours per day, 7 days per week
  Patching 2 hours per day, 7 days per week
- Total: Total of all reporting groups
Arm/Group | Binocular Treatment Younger Cohort (5 to <13 Years) | Patching Treatment Younger Cohort (5 to <13 Years) | Binocular Treatment Older Cohort (13 to <17 Years) | Patching Treatment Older Cohort (13 to <17 Years) | Total
Number analyzed (Participants) | 190 | 195 | 40 | 60 | 485
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 190 | 195 | 40 | 60 | 485
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.4 (1.8) | 8.6 (2.0) | 14.3 (1.1) | 14.3 (1.1) | 9.7 (2.9)
Age, Customized [Count of Participants; unit: Participants]
  Age at enrollment, years : 5 to <7 | 43 | 50 | 0 | 0 | 93
  Age at enrollment, years : 7 to <9 | 78 | 62 | 0 | 0 | 140
  Age at enrollment, years : 9 to <13 | 69 | 83 | 0 | 0 | 152
  Age at enrollment, years : 13 to <17 | 0 | 0 | 40 | 60 | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 89 | 16 | 26 | 229
  Male | 92 | 106 | 24 | 34 | 256
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 134 | 145 | 30 | 43 | 352
  Black/African American | 11 | 12 | 2 | 4 | 29
  Hispanic or Latino | 33 | 24 | 8 | 11 | 76
  Asian, American Indian, Alaskan Native | 9 | 6 | 0 | 1 | 16
  >1 Race | 2 | 5 | 0 | 1 | 8
  Unknown/not reported | 1 | 3 | 0 | 0 | 4
Distance Amblyopic-Eye Visual Acuity [Count of Participants; unit: Participants]
  20/200 (33-37 Letters) | 5 | 4 | 0 | 2 | 11
  20/160 (38-42 Letters) | 6 | 7 | 2 | 5 | 20
  20/125 (43-47 Letters) | 8 | 4 | 4 | 8 | 24
  20/100 (48-52 Letters) | 16 | 12 | 3 | 4 | 35
  20/80 (53-57 Letters) | 30 | 24 | 7 | 12 | 73
  20/63 (58-62 Letters) | 37 | 46 | 6 | 10 | 99
  20/50 (63-67 Letters) | 61 | 52 | 12 | 14 | 139
  20/40 (68-72 Letters) | 27 | 46 | 6 | 5 | 84
Baseline Stereoacuity (Seconds of Arc) [Count of Participants; unit: Participants] — Stereoacuity scores (seconds of arc) were calculated based on the Randot Butterfly (scores: 2000, Nil) and Randot Preschool stereoacuity (scores: 800, 400, 200, 100, 60 and 40) test methods. Lower scores indicate better stereoacuity.
  Results of the Randot Butterfly test were analyzed as 2000 (if correct response). Nil (4000 ) was defined as (1) an incorrect response on the butterfly in absence of a correct response on the 800 seconds of arc level of the Randot Preschool stereoacuity test or (2) an incorrect response on the 800 seconds of arc level if the butterfly was not attempted.
  Participants
    4000 | 69 | 57 | 16 | 29 | 171
    2000 | 28 | 37 | 3 | 7 | 75
    800 | 18 | 26 | 5 | 4 | 53
    400 | 17 | 19 | 7 | 7 | 50
    200 | 23 | 18 | 2 | 4 | 47
    100 | 23 | 23 | 6 | 6 | 58
    60 | 10 | 9 | 1 | 1 | 21
    40 | 2 | 6 | 0 | 2 | 10
Baseline Stereoacuity (Seconds of Arc) [Median (Full Range); unit: Seconds of Arc] — Stereoacuity was tested at near in current refractive correction. Stereoacuity scores (measured as seconds of arc) were calculated based on the Randot Butterfly (scores: 2000, Nil) and Randot Preschool (scores: 800, 400, 200, 100, 60 and 40) stereoacuity test methods as previously described. Lower scores indicate better stereoacuity.
  A logarithm base 10 transformation was used to convert stereoacuity scores (Nil was assigned a score of 4000) to the log scale to calculate descriptive statistics (reported as seconds of arc). Population: Descriptive statistics were computed for baseline stereoacuity by treatment group for all participants and a subset of participants with no history of strabismus.
  The younger (age 5 to <7 years) and older (age 7 to <13 years) were analyzed as separate study cohorts.
  Results of the descriptive analyses are reported as seconds of arc.
  Seconds of Arc
    All participants | 2000 [40 to 4000] | 800 [40 to 4000] | 800 [60 to 4000] | 2000 [40 to 4000] | NA [40 to 4000] — No overall median was calculated because the younger (age 5 to <7 years) and older (age 7 to <13 years) were analyzed as separate age cohorts in effectively separate studies.
    Participants with no history of strabismus: number analyzed (Participants) | 107 | 92 | 22 | 29 | 250
    Participants with no history of strabismus | 400 [40 to 4000] | 400 [40 to 4000] | 400 [60 to 4000] | 800 [60 to 4000] | NA [40 to 4000] — No overall median was calculated because the younger (age 5 to <7 years) and older (age 7 to <13 years) were analyzed as separate age cohorts in effectively separate studies.
Amblyopia Cause [Count of Participants; unit: Participants]
  Strabismus | 22 | 44 | 5 | 9 | 80
  Anisometropia | 107 | 92 | 22 | 29 | 250
  Strabismus/anisometropia combined | 61 | 59 | 13 | 22 | 155

OUTCOME MEASURES:

1. Primary Outcome: Change in Distance Visual Acuity From Baseline in the Younger Cohort (5 to <13 Years)
Description: Monocular distance visual acuity (VA) in current refractive correction (if required) in each eye by a certified examiner using the electronic Amblyopia Treatment Study single-surround HOTV (ATS-HOTV) visual acuity protocol for children <7 years and the Electronic Early Treatment Diabetic Retinoscopy Study (E-ETDRS) visual acuity protocol for children ≥ 7 years on a study-certified acuity tester displaying single surrounded optotypes.
  For the younger cohort, the level of visual acuity is analyzed in the log of the Minimum Angle of Resolution (logMAR) scale (approximate range: -0.2 to 1.7) such that higher scores indicate poorer VA. Change in VA is computed as logMAR lines (positive values indicate improvement), defined as the difference between the enrollment and 16-week acuities (logMAR) multiplied by 10.
Time Frame: Baseline and 16 weeks
Population: Visual acuity analyses included only data from participants who completed the 16-week visit within the predefined analysis window (14 to <20 weeks after randomization), analysis is adjusted for baseline covariates of age and visual acuity.
Measure: Mean (95% Confidence Interval); unit: LogMAR lines
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger
Number analyzed (Participants) | 177 | 186
LogMAR lines
  Adjusted for baseline VA and age | 1.05 [0.85 to 1.24] | 1.35 [1.17 to 1.54]
  Unadjusted | 1.08 [0.86 to 1.29] | 1.32 [1.14 to 1.51]
Statistical Analysis 1: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; The primary outcome measure was change in amblyopic-eye VA from baseline to 16 weeks (14 to <20 week window). The upper limit of a 1-sided 95% confidence interval (CI) was computed on the treatment group difference, using an analysis of covariance (ANCOVA) model, adjusted for baseline age and VA, including only participants completing the 16-week outcome in a modified intent-to-treat analysis. There was no imputation for missing data; Test type: Non-Inferiority — Our sample size was computed to have 90% power with a type I error of 5% for a non-inferiority limit of 0.05 logMAR (0.5 lines), assuming a standard deviation of change of 0.15 logMAR (1.5 lines) based on prior Pediatric Eye Disease Investigator Group (PEDIG) studies, and no more than 10% loss to follow-up; Mean Difference (Final Values) = 0.31, 95% CI 1-sided [upper limit 0.53] — A 1-sided upper 95% confidence interval was computed on the adjusted group difference (patching - binocular treatment) evaluating change in amblyopic-eye visual acuity from baseline to the 16-week visit. Positive values favor the patching group
Statistical Analysis 2: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; The primary analysis was repeated for the treatment group comparison of change in amblyopic-eye VA from baseline to 16 weeks, adjusting for baseline covariates of age and visual acuity. For this sensitivity analysis, the primary analysis repeated but excluded data from participants (n=35) who completed the 16-week visit outside of the pre-defined protocol window (16 +/- 1 week); Test type: Non-Inferiority — Our sample size was computed to have 90% power with a type I error of 5% for a non-inferiority limit of 0.05 logMAR (0.5 lines), assuming a standard deviation of change of 0.15 logMAR (1.5 lines) based on prior PEDIG studies, and no more than 10% loss to follow-up; Mean Difference (Final Values) = 0.30, 95% CI 1-sided [upper limit 0.53] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; The primary analysis was repeated for the treatment group comparison of change in amblyopic-eye from baseline to 16 weeks, adjusting for baseline covariates of age and visual acuity. For this sensitivity analysis, multiple imputation was used to impute 16-week visual acuity scores for participants who missed the exam (n=15) or completed the 16-week exam outside of the pre-specified analysis window (n=7); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Mean Difference (Final Values) = 0.31, 95% CI 1-sided [upper limit 0.54] — A 1-sided 95% confidence interval was computed on the adjusted group difference (patching - binocular treatment) evaluating change in amblyopic-eye visual acuity from baseline to the 16-week visit. Positive values favor the patching group
Statistical Analysis 4: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; The primary analysis was repeated for the treatment group comparison of change in amblyopic-eye VA from baseline to 16 weeks, adjusting for baseline covariates for age and visual acuity. For this post hoc sensitivity analysis, all participants with 16-week exams were included in the analysis regardless of whether or not the exam was completed within the pre-specified analysis window (14 to <20 weeks after randomization); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Mean Difference (Final Values) = 0.33, 95% CI 1-sided [upper limit 0.56] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; The primary analysis was repeated for the treatment group comparison of change in amblyopic-eye VA from baseline to 16-weeks, adjusting for baseline covariates of age and visual acuity. For this sensitivity analysis, we excluded 16-week outcomes from enrolled participants who were subsequently found to be ineligible for the study (n=7); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Mean Difference (Final Values) = 0.30, 95% CI 1-sided [upper limit 0.53] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; The primary analysis was repeated for the treatment group comparison of change in amblyopic-eye visual acuity from baseline to 16 week, adjusting for baseline covariates of age and visual acuity. For this sensitivity analysis, we excluded 16-week outcomes from participants who received alternative treatment for at least 1 week during study follow-up (n=4); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Mean Difference (Final Values) = 0.33, 95% CI 1-sided [upper limit 0.55] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 7: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; Analysis of covariance included baseline age and visual acuity as adjustment covariates. The primary outcome measure was change in amblyopic-eye VA from baseline to 16 weeks (14 to <20 week window). For this post hoc analysis, a 2-sided 95% confidence interval (CI) was computed on the treatment group difference, using an analysis of covariance (ANCOVA) model, adjusted for baseline age and VA, including only participants completing the 16-week outcome in a modified intent-to-treat analysis; Test type: Superiority; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [0.04 to 0.58] — A 2-sided 95% confidence interval was computed on the adjusted treatment group difference evaluating change in amblyopic-eye visual acuity from baseline to the 16-week visit. Positive estimate values favor the patching treatment group

2. Primary Outcome: Mean Amblyopic Eye Visual Acuity (Younger Cohort)
Description: Monocular distance visual acuity (VA) in current refractive correction (if required) in each eye by a certified examiner using the electronic Amblyopia Treatment Study single-surround HOTV (ATS-HOTV) visual acuity protocol for children <7 years and the Electronic Early Treatment Diabetic Retinoscopy Study (E-ETDRS) visual acuity protocol for children ≥ 7 years on a study-certified acuity tester displaying single surrounded optotypes.
  For the younger cohort, the level of visual acuity is analyzed in the log of the Minimum Angle of Resolution (logMAR) scale (approximate range: -0.2 to 1.7) such that higher scores indicate poorer VA.
Time Frame: 16 Weeks from baseline
Population: Visual acuity analyses included only data from participants who completed the 16-week visit within the predefined analysis window (14 to <20 weeks after randomization).
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger
Number analyzed (Participants) | 177 | 186
LogMAR | 0.41 (0.21) | 0.35 (0.20)

3. Primary Outcome: Mean Change in Amblyopic-eye Visual Acuity in the Older Cohort (13 to <17 Years)
Description: Monocular distance visual acuity (VA) in current refractive correction (if required) in each eye by a certified examiner using the Electronic Early Treatment Diabetic Retinoscopy Study (E-ETDRS) visual acuity protocol for children ≥ 7 years on a study-certified acuity tester displaying single surrounded optotypes.
  For the analyses in the older cohort, the level of VA is measured as letter scores (approximate range: 0 to 97 letters, lower scores indicate poorer VA) and change in VA from baseline is measured in letters (positive values indicate improvement), defined as the difference in letter scores between enrollment and follow-up.
Time Frame: Baseline and 16 weeks
Population: Mean change in amblyopic-eye visual acuity from baseline to 16 weeks from participants who completed 16-week visit within pre-specified analysis window (148 to 196 days after randomization)
Measure: Mean (95% Confidence Interval); unit: letters
Groups:
- Binocular Treatment Older: Age 13 to <17
  Binocular computer game play 1 hour per day, 7 days per week (minimum of 4 days per week)
  iPad®: Binocular therapy on iPad®
- Patching Treatment Older: Age 13 to <17
  Patching 2 hours per day, 7 days per week
  Patching 2 hours per day, 7 days per week
Arm/Group | Binocular Treatment Older | Patching Treatment Older
Number analyzed (Participants) | 39 | 56
letters
  Unadjusted | 3.5 [1.3 to 5.7] | 6.5 [4.4 to 8.5]
  Adjusted for baseline visual acuity | 3.7 [1.3 to 6.0] | 6.3 [4.4 to 8.3]
Statistical Analysis 1: Comparison: Binocular Treatment Older vs Patching Treatment Older; A modified intent-to-treat analysis was performed using an ANCOVA model to compare the effectiveness of two treatments (2-sided hypothesis test), adjusting for baseline visual acuity. The primary outcome measure was change in amblyopic-eye VA from baseline to 16 weeks (14 to <20 week window). A 2-sided 95% confidence interval (CI) was computed on the adjusted treatment group difference at 16 weeks. There was no imputation for missing data; Test type: Superiority; p = 0.082, ANCOVA — a priori threshold for statistical significance: 2-sided type I error rate of 5%; Adjusted for baseline amblyopic-eye visual acuity; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-5.7 to 0.3] — A 2-sided 95% confidence interval was computed on the adjusted treatment group difference (binocular treatment - patching) evaluating change in amblyopic-eye visual acuity from baseline to the 16-week visit
Statistical Analysis 2: Comparison: Binocular Treatment Older vs Patching Treatment Older; A modified intent-to-treat analysis was performed using an ANCOVA model to compare the change in amblyopic-eye visual acuity from baseline to 16 weeks for two treatments (2-sided hypothesis test), adjusting for baseline visual acuity. For this sensitivity analyses, the primary analysis was repeated but excluded data from participants who completed the 16-week visit outside of the pre-specified 16 +/- 1 week protocol window (n=10 participants); Test type: Superiority; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-5.9 to 0.5] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Binocular Treatment Older vs Patching Treatment Older; A modified intent-to-treat analysis was performed using an ANCOVA model to compare the change in amblyopic-eye visual acuity from baseline to 16 weeks (14 to <20 week window) for two treatments (2-sided hypothesis test), adjusting for baseline visual acuity. For this sensitivity analyses, the primary analysis was repeated but excluded data from participants later found to be ineligible for the study (n=2); Test type: Superiority; Mean Difference (Final Values) = -2.8, 95% CI 2-sided [-5.9 to 0.3] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Binocular Treatment Older vs Patching Treatment Older; The primary analysis was repeated for the treatment group comparison of change in amblyopic-eye from baseline to 16 weeks, adjusting for baseline visual acuity. For this sensitivity analysis, multiple imputation was used to impute 16-week visual acuity scores for participants who missed the exam (n=3) or completed the 16-week exam outside of the pre-specified analysis window (n=2); Test type: Superiority; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-5.0 to 1.2] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Binocular Treatment Older vs Patching Treatment Older; An ANCOVA model was fit to compare the change in amblyopic-eye visual acuity from baseline to 16 weeks (14 to <20 week window) for two treatments (2-sided hypothesis test), adjusting for baseline visual acuity. For this post hoc sensitivity analyses, the primary analysis was repeated but included data from participants who completed the 16-week visit outside the analysis window (n=2, range:14 to 28 weeks post randomization); Test type: Superiority; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-5.5 to 0.5] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Binocular Treatment Older vs Patching Treatment Older; An ANCOVA model was fit to compare the change in amblyopic-eye visual acuity from baseline to 16 weeks (14 to <20 week window) for two treatments (2-sided hypothesis test), adjusting for baseline visual acuity. For this sensitivity analyses, the primary analysis was repeated but included prior amblyopia treatment as an adjustment covariate (in addition to baseline visual acuity) in the model; Test type: Superiority; Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-5.7 to 0.4] — [estimate comment as in outcome 3, analysis 1]

4. Primary Outcome: Mean Amblyopic-eye Visual Acuity in the Older Cohort (13 to <17 Years)
Description: as for outcome 3
Time Frame: 16 weeks
Population: Participants that completed 16-week visit within pre-specified analysis window (148 to 196 days after randomization)
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Binocular Treatment Older | Patching Treatment Older
Number analyzed (Participants) | 39 | 56
letters | 62.0 (9.7) | 62.5 (11.6)

5. Primary Outcome: Distribution of Change in Amblyopic-eye Visual Acuity
Description: Monocular distance visual acuity (VA) in current refractive correction (if required) in each eye by a certified examiner using the electronic Amblyopia Treatment Study single-surround HOTV (ATS-HOTV) visual acuity protocol for children <7 years and the Electronic Early Treatment Diabetic Retinoscopy Study (E-ETDRS) visual acuity protocol for children ≥ 7 years on a study-certified acuity tester displaying single surrounded optotypes.
  Younger cohort: The level of VA is analyzed in the log of the Minimum Angle of Resolution (logMAR) scale (previously defined) and change in VA from baseline as logMAR lines (previously defined).
  Older cohort: The level of VA is measured as letter scores (previously defined) and VA change from baseline is measured in letters (previously defined).
Time Frame: Baseline and 16 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Binocular Treatment Older Cohort: Binocular computer game play 1 hour per day, 7 days per week (minimum of 4 days per week)
  iPad®: Binocular therapy on iPad®
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger | Binocular Treatment Older Cohort | Patching Treatment Older
Number analyzed (Participants) | 177 | 186 | 39 | 56
Participants
  ≥ 3 LogMAR lines (≥ 15 letters) better | 19 | 29 | 2 | 7
  2 LogMAR lines (10-14 letters) better | 32 | 36 | 4 | 10
  1 LogMAR line (5-9 letters) better | 47 | 46 | 9 | 19
  0 LogMAR line (within 4 letters) | 64 | 69 | 22 | 18
  1 LogMAR line (5-9 letters) worse | 12 | 6 | 1 | 1
  2 LogMAR lines (10-14 letters) worse | 1 | 0 | 0 | 0
  ≥3 LogMAR lines (≥ 15 letters) worse | 2 | 0 | 1 | 1

6. Primary Outcome: Distribution of Amblyopic-eye Visual Acuity
Description: as for outcome 5
Time Frame: At 16 weeks
Population: Participants that completed 16-week visit within pre-specified analysis window (148 to 196 days after randomization)
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger | Binocular Treatment Older | Patching Treatment Older
Number analyzed (Participants) | 177 | 186 | 39 | 56
Participants
  20/200 (33-37 letters) | 2 | 1 | 1 | 1
  20/160 (38-42 letters) | 2 | 3 | 0 | 1
  20/125 (43-47 letters) | 10 | 2 | 2 | 4
  20/100 (48-52 letters) | 12 | 7 | 4 | 7
  20/80 (53-57 letters) | 18 | 17 | 5 | 8
  20/63 (58-62 letters) | 25 | 22 | 5 | 4
  20/50 (63-67 letters) | 30 | 38 | 11 | 9
  20/40 (68-72 letters) | 32 | 37 | 6 | 7
  20/32 (73-77 letters) | 33 | 27 | 4 | 11
  20/25 (78-82 letters) | 8 | 22 | 0 | 3
  20/20 (83-87 letters) | 3 | 10 | 1 | 1
  20/16 (88-92 letters) | 2 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Amblyopic-eye VA Improvement of 2 or More logMAR Lines (10 or More Letters if E-ETDRS) From Baseline
Description: as for outcome 5
Time Frame: Baseline and 16-week visit
Population: Analysis was limited to participants who completed the 16-week visit within the pre-specified analysis window (14 to <20 weeks after randomization).
Measure: Count of Participants; unit: Participants
Groups:
- Patching Treatment Older Cohort: Patching 2 hours per day, 7 days per week
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger | Binocular Treatment Older Cohort | Patching Treatment Older Cohort
Number analyzed (Participants) | 177 | 186 | 39 | 56
Participants | 51 | 65 | 6 | 17
Statistical Analysis 1: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; Binomial regression was used for the treatment group comparison of the proportion of participants classified as improving 2 or more logMAR lines (10 or more letters if E-ETDRS) from baseline at the 16-week visit, adjusting for baseline age group (5 to <7, 7 to <13 years) and baseline visual acuity (treated as a continuous covariate); Test type: Superiority; Risk Difference (RD) = 5, 95% CI 2-sided [-4 to 13] — Binomial regression was used to compare the group proportions (patching - binocular treatment) of participants classified as improving 2 or more logMAR lines from baseline at the 16-week visit
Statistical Analysis 2: Comparison: Binocular Treatment Older Cohort vs Patching Treatment Older Cohort; Binomial regression was used for the treatment group comparison of the proportion of participants classified as improving 2 or more logMAR lines (10 or more letters if E-ETDRS) from baseline at the 16-week visit, adjusting for baseline visual acuity; Test type: Superiority; Risk Difference (RD) = -15, 95% CI 2-sided [-31 to 2] — Binomial regression was used to compare the group proportions (binocular treatment - patching) of participants classified as improving 2 or more logMAR lines (≥ 10 letters) from baseline at the 16-week visit

8. Secondary Outcome: Number of Participants With Resolution of Amblyopia
Description: Monocular distance visual acuity (VA) in current refractive correction (if required) in each eye by a certified examiner using the electronic Amblyopia Treatment Study single-surround HOTV (ATS-HOTV) visual acuity protocol for children <7 years and the Electronic Early Treatment Diabetic Retinoscopy Study (E-ETDRS) visual acuity protocol for children ≥ 7 years on a study-certified acuity tester displaying single surrounded optotypes.
  The level of VA is analyzed in the log of the Minimum Angle of Resolution (logMAR) scale (previously defined) for the younger cohort and as letter scores (previously defined) for the older cohort.
  Resolution of amblyopia was defined as having an amblyopic-eye VA of 20/25 or better (≥ 78 letters if E-ETDRS) and within 1 logMAR line (5 letters if E-ETDRS) of the fellow eye VA.
Time Frame: 16-week visit
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger | Binocular Treatment Older Cohort | Patching Treatment Older Cohort
Number analyzed (Participants) | 177 | 186 | 39 | 56
Participants | 8 | 18 | 0 | 0
Statistical Analysis 1: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; Binomial regression was used for the treatment group comparison of the proportion of participants classified as improving 2 or more logMAR lines (10 or more letters if E-ETDRS) from baseline at the 16-week visit, adjusting for baseline age group (5 to <7, 7 to <13 years) and baseline visual acuity (20/40, 20/50 or worse); Test type: Superiority; Risk Difference (RD) = 2, 95% CI 2-sided [-1 to 5] — Binomial regression was used to compare the group proportions (patching - binocular treatment) of participants classified as having amblyopia resolution at the 16-week visit

9. Secondary Outcome: Time Course of Visual Acuity Improvement
Description: Monocular distance visual acuity (VA) in current refractive correction (if required) in each eye by a certified examiner using the electronic Amblyopia Treatment Study single-surround HOTV (ATS-HOTV) visual acuity protocol for children <7 years and the Electronic Early Treatment Diabetic Retinoscopy Study (E-ETDRS) visual acuity protocol for children ≥ 7 years on a study-certified acuity tester displaying single surrounded optotypes.
  For the younger cohort, the level of VA is analyzed in the log of the Minimum Angle of Resolution (logMAR) scale (approximate range: -0.2 to 1.7, higher values indicate poorer VA) and change in VA from baseline as logMAR lines (positive values indicate improvement), defined as the difference between the enrollment and follow-up acuities (logMAR) multiplied by 10.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks and 16 weeks
Population: Analysis included participants with at least one follow-up visit (completed within the analysis window). There were 6 participants (4 in the binocular group, 2 in the patching group) who were excluded from the time course analysis because they did not have any follow-up exams.
Measure: Mean (Standard Deviation); unit: logMAR lines
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger
Number analyzed (Participants) | 186 | 193
logMAR lines
  4-week visit: number analyzed (Participants) | 176 | 188
  4-week visit | 0.53 (1.14) | 0.76 (1.09)
  8-week visit: number analyzed (Participants) | 172 | 186
  8-week visit | 0.76 (1.18) | 1.03 (1.23)
  12-week visit: number analyzed (Participants) | 178 | 187
  12-week visit | 0.90 (1.37) | 1.21 (1.26)
  16-week visit: number analyzed (Participants) | 177 | 186
  16-week visit | 1.08 (1.45) | 1.32 (1.26)
Statistical Analysis 1: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; A linear mixed model was used to compare the rate of amblyopic-eye visual acuity improvement between the treatment groups. The ANCOVA model included an interaction term with treatment group and time to compare the change in visual acuity over follow-up by treatment group, adjusting for the main effects of the interaction term and baseline covariates of age and visual acuity. If the interaction term was not statistically significant (p>0.05), no further comparisons would be performed; Test type: Superiority; p = 0.83, ANCOVA — For testing the interaction term, the a priori threshold for statistical significance was 0.05; Previously described above in the Statistical Analysis Overview section

10. Secondary Outcome: Younger Cohort: Change in Distance Visual Acuity From Baseline According to Subgroups
Description: Monocular distance visual acuity (VA) in current refractive correction (if required) in each eye by a certified examiner using the electronic Amblyopia Treatment Study single-surround HOTV (ATS-HOTV) visual acuity protocol for children <7 years and the Electronic Early Treatment Diabetic Retinoscopy Study (E-ETDRS) visual acuity protocol for children ≥ 7 years on a study-certified acuity tester displaying single surrounded optotypes.
  For the younger cohort, the level of VA is analyzed in the log of the Minimum Angle of Resolution (logMAR) scale (previously defined) and change in VA from baseline as logMAR lines (previously defined, positive values indicate improvement), For both descriptive and formal subgroup analyses, all subgroup factors were pre-specified except for baseline stereoacuity (nil, better than nil). We performed post hoc descriptive analyses to explore treatment effect by baseline age (5 to <7 yrs, 7 to <13 yrs) and prior amblyopia treatment (yes/no).
Time Frame: Baseline and 16 weeks
Population: Visual acuity analyses included only data from participants who completed the 16-week visit within the predefined analysis window (14 to <20 weeks after randomization). Formal subgroup analyses are adjusted for baseline covariates of visual acuity and age.
Measure: Mean (Standard Deviation); unit: LogMAR lines
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger
Number analyzed (Participants) | 177 | 186
LogMAR lines
  Female: number analyzed (Participants) | 89 | 83
  Female | 1.2 (1.5) | 1.4 (1.2)
  Male: number analyzed (Participants) | 88 | 103
  Male | 1.0 (1.4) | 1.3 (1.3)
  White/Non-Hispanic: number analyzed (Participants) | 122 | 139
  White/Non-Hispanic | 1.0 (1.5) | 1.3 (1.2)
  Non-White or Hispanic: number analyzed (Participants) | 54 | 44
  Non-White or Hispanic | 1.2 (1.5) | 1.3 (1.4)
  Age at baseline: 5 to <7 years: number analyzed (Participants) | 39 | 49
  Age at baseline: 5 to <7 years | 1.9 (1.8) | 2.0 (1.4)
  Age at baseline: 7 to <13 years: number analyzed (Participants) | 138 | 137
  Age at baseline: 7 to <13 years | 0.8 (1.2) | 1.1 (1.1)
  Baseline amblyopic-eye VA: 20/80 to 20/200: number analyzed (Participants) | 64 | 50
  Baseline amblyopic-eye VA: 20/80 to 20/200 | 1.1 (1.6) | 1.3 (1.3)
  Baseline amblyopic-eye VA: 20/63: number analyzed (Participants) | 32 | 45
  Baseline amblyopic-eye VA: 20/63 | 1.3 (1.6) | 1.4 (1.3)
  Baseline amblyopic-eye VA: 20/50: number analyzed (Participants) | 55 | 50
  Baseline amblyopic-eye VA: 20/50 | 1.0 (1.3) | 1.3 (1.3)
  Baseline amblyopic-eye VA: 20/40: number analyzed (Participants) | 26 | 41
  Baseline amblyopic-eye VA: 20/40 | 0.8 (1.2) | 1.2 (1.2)
  Baseline stereoacuity: Nil: number analyzed (Participants) | 68 | 55
  Baseline stereoacuity: Nil | 0.7 (1.3) | 1.1 (1.1)
  Baseline stereoacuity: Better than Nil: number analyzed (Participants) | 109 | 131
  Baseline stereoacuity: Better than Nil | 1.3 (1.5) | 1.4 (1.3)
  No presence of a near heterotropia at baseline: number analyzed (Participants) | 122 | 117
  No presence of a near heterotropia at baseline | 1.1 (1.3) | 1.3 (1.2)
  Presence of a near heterotropia at baseline: number analyzed (Participants) | 55 | 69
  Presence of a near heterotropia at baseline | 0.9 (1.7) | 1.4 (1.3)
  No prior amblyopia treatment: number analyzed (Participants) | 41 | 39
  No prior amblyopia treatment | 1.9 (1.5) | 2.2 (1.3)
  Prior amblyopia treatment: number analyzed (Participants) | 136 | 147
  Prior amblyopia treatment | 0.8 (1.4) | 1.1 (1.2)
  Baseline: Age 5 to <7 yrs, no prior treatment: number analyzed (Participants) | 19 | 19
  Baseline: Age 5 to <7 yrs, no prior treatment | 2.5 (1.5) | 2.8 (0.8)
  Baseline: Age 5 to <7 yrs, prior treatment: number analyzed (Participants) | 20 | 30
  Baseline: Age 5 to <7 yrs, prior treatment | 1.4 (1.9) | 1.4 (1.4)
  Baseline: Age 7 to <13 yrs, no prior treatment: number analyzed (Participants) | 22 | 20
  Baseline: Age 7 to <13 yrs, no prior treatment | 1.3 (1.2) | 1.5 (1.3)
  Baseline: Age 7 to <13 yrs, prior treatment: number analyzed (Participants) | 116 | 117
  Baseline: Age 7 to <13 yrs, prior treatment | 0.7 (1.2) | 1.0 (1.1)
Statistical Analysis 1: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; Exploratory subgroup analyses were conducted to assess the treatment effect according to subgroups of baseline factors. An analysis of covariance was used to test the interaction between treatment group and gender, adjusting for the main effects of the interaction term and baseline covariates of age and visual acuity; Test type: Superiority; p = 0.83, ANCOVA — The a priori threshold for statistical significance of the interaction term (gender and treatment group) was 0.05; Previously described in the Statistical Analysis Overview
Statistical Analysis 2: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; Exploratory subgroup analyses were conducted to assess the treatment effect according to subgroups of baseline factors. An analysis of covariance was used to test the interaction between treatment group and race/ethnicity status (White/non-Hispanic, Non-White or Hispanic), adjusting for the main effects of the interaction term and baseline covariates of age and visual acuity; Test type: Superiority; p = 0.54, ANCOVA — The a priori threshold for statistical significance of the interaction term (race/ethnicity status and treatment group) was 0.05; Four participants (1 binocular treatment group, 3 patching group) were excluded from the analysis due to unknown/not reported race/ethnicity status
Statistical Analysis 3: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; Exploratory subgroup analyses were conducted to assess the treatment effect according to subgroups of baseline factors. An analysis of covariance was used to test the interaction between treatment group and age at baseline (treated as a continuous factor in the model), adjusting for the main effects of the interaction term and baseline visual acuity; Test type: Superiority; p = 0.80, ANCOVA — The a priori threshold for statistical significance of the interaction term (age and treatment group) was 0.05
Statistical Analysis 4: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; Exploratory subgroup analyses were conducted to assess the treatment effect according to subgroups of baseline factors. An analysis of covariance was used to test the interaction between treatment group and baseline amblyopic-eye visual acuity (treated as a continuous factor in the model), adjusting for the main effects of the interaction term and baseline age; Test type: Superiority; p = 0.99, ANCOVA — The a priori threshold for statistical significance of the interaction term (baseline amblyopic-eye visual acuity and treatment group) was 0.05
Statistical Analysis 5: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; Exploratory subgroup analyses were conducted to assess the treatment effect according to subgroups of baseline factors. An analysis of covariance was used to test the interaction between treatment group and prior amblyopia treatment (Yes/No), adjusting for the main effects of the interaction term and baseline covariates of age and visual acuity; Test type: Superiority; p = 0.87, ANCOVA — The a priori threshold for statistical significance of the interaction term (prior amblyopia treatment and treatment group) was 0.05
Statistical Analysis 6: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; Exploratory subgroup analyses were conducted to assess the treatment effect according to subgroups of baseline factors. An analysis of covariance was used to test the interaction between treatment group and baseline stereoacuity (nil, better than nil), adjusting for the main effects of the interaction term and baseline covariates of age and visual acuity; Test type: Superiority; p = 0.33, ANCOVA — The a priori threshold for statistical significance of the interaction term (baseline stereoacuity and treatment group) was 0.05
Statistical Analysis 7: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; Exploratory subgroup analyses were conducted to assess the treatment effect according to subgroups of baseline factors. An analysis of covariance was used to test the interaction between treatment group and presence of a near heterotropia (measured by SPCT) at baseline (Yes/No), adjusting for the main effects of the interaction term and baseline covariates of age and visual acuity; Test type: Superiority; p = 0.23, ANCOVA — The a priori threshold for statistical significance of the interaction term (presence of a near heterotropia at baseline and treatment group) was 0.05

11. Secondary Outcome: Older Cohort: Change in Distance Visual Acuity From Baseline According to Subgroups
Description: Monocular distance visual acuity (VA) in current refractive correction (if required) in each eye by a certified examiner using the Electronic Early Treatment Diabetic Retinoscopy Study (E-ETDRS) visual acuity protocol for children ≥ 7 years on a study-certified acuity tester displaying single surrounded optotypes.
  For the analyses in the older cohort, the level of VA is measured as letter scores (previously defined) and change in VA from baseline is measured in letters (positive values indicate improvement), defined as the difference in letter scores between enrollment and follow-up.
  Subgroup factors of interest were pre-specified except for baseline stereoacuity (nil, better than nil).
Time Frame: Baseline and 16 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Binocular Treatment Older Cohort | Patching Treatment Older Cohort
Number analyzed (Participants) | 39 | 56
Letters
  Female | 1.0 (6.8) | 6.0 (6.7)
  Male | 5.0 (6.4) | 6.8 (8.4)
  White/Non-Hispanic | 3.6 (7.1) | 6.4 (7.6)
  Non-White or Hispanic | 3.2 (6.1) | 6.7 (8.2)
  Baseline amblyopic-eye VA: 20/80 to 20/200 | 5.2 (7.8) | 7.1 (8.3)
  Baseline amblyopic-eye VA: 20/63 | 3.2 (2.8) | 5.0 (10.6)
  Baseline amblyopic-eye VA: 20/50 | 2.9 (4.2) | 6.0 (4.4)
  Baseline amblyopic-eye VA: 20/40 | -0.4 (10.9) | 6.8 (6.4)
  No prior amblyopia treatment | 2.9 (6.4) | 10.3 (8.0)
  Prior amblyopia treatment | 3.6 (7.0) | 6.0 (7.6)
  Baseline stereoacuity: Nil | 4.1 (7.7) | 5.7 (7.6)
  Baseline stereoacuity: Better than Nil | 3.0 (6.2) | 7.2 (7.8)
  No presence of a near heterotropia at baseline | 2.0 (6.1) | 5.6 (8.1)
  Presence of a near heterotropia at baseline | 5.7 (7.4) | 7.9 (6.9)

12. Secondary Outcome: Distribution of Stereoacuity Scores
Description: Stereoacuity was tested at near in current refractive correction. Stereoacuity scores (measure as seconds of arc) were calculated based on the Randot Butterfly (scores: 2000, Nil) and Randot Preschool stereoacuity (scores: 800, 400, 200, 100, 60 and 40) test methods.
  Lower scores indicate better stereoacuity. Results of the Randot Butterfly test were analyzed as 2000 seconds of arc (if correct response). Nil was assigned a score of 4000 seconds of arc and was defined as (1) an incorrect response on the butterfly in absence of a correct response on the 800 seconds of arc level of the Randot Preschool stereoacuity test or (2) an incorrect response on the 800 seconds of arc level if the butterfly was not attempted.
Time Frame: 16 weeks
Population: The analysis included all participants who completed a 16-week exam regardless of whether or not the exam was completed within the pre-specified analysis window.
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger | Binocular Treatment Older Cohort | Patching Treatment Older Cohort
Number analyzed (Participants) | 182 | 188 | 39 | 58
Participants
  Missing/Not done | 1 | 0 | 0 | 0
  4000 seconds of arc | 62 | 50 | 13 | 25
  2000 seconds of arc | 32 | 32 | 6 | 11
  800 seconds of arc | 19 | 28 | 6 | 7
  400 seconds of arc | 14 | 17 | 3 | 4
  200 seconds of arc | 15 | 27 | 2 | 2
  100 seconds of arc | 17 | 19 | 6 | 2
  60 seconds of arc | 10 | 11 | 2 | 2
  40 seconds of arc | 12 | 4 | 1 | 5

13. Secondary Outcome: Median Stereoacuity Score (Seconds of Arc)
Description: Stereoacuity was tested at near in current refractive correction. Stereoacuity scores (measure as seconds of arc) were calculated based on the Randot Butterfly (scores: 2000, Nil) and Randot Preschool stereoacuity (scores: 800, 400, 200, 100, 60 and 40) test methods. Lower scores indicate better stereoacuity.
  Results of the Randot Butterfly test were analyzed as 2000 seconds of arc (if correct response). Nil was assigned a score of 4000 seconds of arc and was defined as (1) an incorrect response on the butterfly in absence of a correct response on the 800 seconds of arc level of the Randot Preschool stereoacuity test or (2) an incorrect response on the 800 seconds of arc level if the butterfly was not attempted.
  A logarithm base 10 transformation was used to convert stereoacuity scores (seconds of arc) to the log scale (conversion reference listed below), which was used to calculate descriptive statistics. Results of the descriptive analyses are reported as seconds of arc.
Time Frame: 16 weeks
Population: Participants who completed stereoacuity testing at the 16-week visit (regardless of whether or not the visit was completed within the pre-specified analysis window).
  Descriptive analyses were repeated for a subset of participants with no history of strabismus.
Measure: Median (Full Range); unit: Seconds of arc
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger | Binocular Treatment Older Cohort | Patching Treatment Older Cohort
Number analyzed (Participants) | 181 | 188 | 39 | 58
Seconds of arc
  All participants | 2000 [40 to 4000] | 800 [40 to 4000] | 800 [40 to 4000] | 2000 [40 to 4000]
  Participants with no history of strabismus: number analyzed (Participants) | 104 | 90 | 27 | 21
  Participants with no history of strabismus | 400 [40 to 4000] | 400 [40 to 4000] | 400 [40 to 4000] | 2000 [40 to 4000]

14. Secondary Outcome: Distribution of Stereoacuity Scores (Participants With no History of Strabismus)
Description: as for outcome 12
Time Frame: 16 weeks
Population: The analysis was limited to a subset of participants (no history of strabismus) who completed a 16-week exam regardless of whether or not the exam was completed within the pre-specified analysis window.
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger | Binocular Treatment Older Cohort | Patching Treatment Older Cohort
Number analyzed (Participants) | 105 | 90 | 21 | 27
Participants
  Missing/Not done | 1 | 0 | 0 | 0
  4000 seconds of arc | 23 | 13 | 4 | 10
  2000 seconds of arc | 14 | 12 | 1 | 4
  800 seconds of arc | 12 | 14 | 4 | 3
  400 seconds of arc | 10 | 10 | 2 | 1
  200 seconds of arc | 12 | 17 | 2 | 1
  100 seconds of arc | 14 | 15 | 5 | 1
  60 seconds of arc | 9 | 6 | 2 | 2
  40 seconds of arc | 10 | 3 | 1 | 5

15. Secondary Outcome: Distribution of Change in Stereoacuity Scores From Baseline
Description: Stereoacuity was tested at near in current refractive correction. Stereoacuity scores (seconds of arc) were calculated based on the Randot Butterfly (scores: 2000, Nil) and Randot Preschool stereoacuity (scores: 800, 400, 200, 100, 60 and 40) test methods. Lower scores indicate better stereoacuity.
  Results of the Randot Butterfly test were analyzed as 2000 (if correct response). Nil (4000 ) was defined as (1) an incorrect response on the butterfly in absence of a correct response on the 800 seconds of arc level of the Randot Preschool stereoacuity test or (2) an incorrect response on the 800 seconds of arc level if the butterfly was not attempted.
  For each visit, stereoacuity scores were ordered and assigned a rank score. Change in stereoacuity was calculated as the difference in ranked score between the enrollment and 16-week stereoacuity scores.
Time Frame: Baseline and 16 weeks
Population: The analysis included all participants who completed stereoacuity testing at both baseline and the 16-week visit (regardless of whether or not the exam was completed within the pre-specified analysis window).
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger | Binocular Treatment Older Cohort | Patching Treatment Older Cohort
Number analyzed (Participants) | 181 | 188 | 39 | 58
Participants
  2 or more levels worse | 19 | 24 | 4 | 8
  Within 1 level | 130 | 122 | 29 | 38
  2 or more levels better | 32 | 42 | 6 | 12
Statistical Analysis 1: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; The Wilcoxon rank-sum test was used to compare the distribution of change in stereoacuity levels from baseline to 16 weeks by treatment group; Test type: Superiority; p = 0.66, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was 0.05
Statistical Analysis 2: Comparison: Binocular Treatment Older Cohort vs Patching Treatment Older Cohort; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p = 0.83, Wilcoxon (Mann-Whitney) — A priori threshold for statistical significance was 0.05

16. Secondary Outcome: Distribution of Change in Stereoacuity Scores From Baseline (Participants With no History of Strabismus)
Description: as for outcome 15
Time Frame: Baseline and 16 weeks
Population: The analysis included a subset of participants with no history of strabismus who completed stereoacuity testing at both baseline and the 16-week visit (regardless of whether or not the exam was completed within the pre-specified analysis window).
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger | Binocular Treatment Older Cohort | Patching Treatment Older Cohort
Number analyzed (Participants) | 104 | 90 | 21 | 27
Participants
  2 or more levels worse | 12 | 14 | 2 | 4
  Within 1 level | 67 | 58 | 15 | 16
  2 or more levels better | 25 | 18 | 4 | 7
Statistical Analysis 1: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p = 0.19, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was 0.05
Statistical Analysis 2: Comparison: Binocular Treatment Older Cohort vs Patching Treatment Older Cohort; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p = 0.69, Wilcoxon (Mann-Whitney) — A priori threshold for statistical significance was 0.05

17. Secondary Outcome: Binocular Treatment Group: Adherence and Fellow-eye Contrast (iPad Log File Data)
Description: Participants assigned to binocular treatment were prescribed the binocular falling blocks game for 1 hour per day (allowing division into shorter sessions), 7 days per week for 16 weeks, with instructions to perform therapy a minimum of 4 days per week if unable to play for 7 days per week.
  The iPad device automatically recorded duration of game play, fellow-eye contrast, and performance. Adherence was calculated as the total hours of game play since baseline divided by the total prescribed hours (based on intended dose of 1 hour a day, 7 days per week) since baseline.
  The fellow-eye contrast was initially set to 20% (amblyopic eye always at 100%) and automatically increased or decreased by 10% increments (lowest level of 10%) or left unchanged from the last contrast level, based on the previous day's game play duration (at least 30 minutes required for contrast change) and performance (increased if scored 1000 points or more).
  Post hoc analysis: 4-week fellow-eye contrast.
Time Frame: Entire study period, up to 16 weeks
Population: The descriptive analysis included data from participants in the binocular treatment group who had log file data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Treatment Younger | Binocular Treatment Older Cohort
Number analyzed (Participants) | 176 | 38
Participants
  Completed >75% prescribed game play | 39 | 5
  Fellow-eye contrast of 100% (16 weeks) | 86 | 23
  Fellow-eye contrast of 20% or worse (16 weeks) | 31 | 3
  Fellow-eye contrast of 100% (4 weeks): number analyzed (Participants) | 173 | 36
  Fellow-eye contrast of 100% (4 weeks) | 35 | 6

18. Secondary Outcome: Binocular Treatment Group: Median Adherence With Prescribed Game Play (iPad Log File Data)
Description: Participants assigned to binocular treatment were prescribed the binocular falling blocks game for 1 hour per day (allowing division into shorter sessions), 7 days per week for 16 weeks, with instructions to perform therapy a minimum of 4 days per week if unable to play for 7 days per week.
  The iPad device automatically recorded duration of game play, fellow-eye contrast, and performance.
  Adherence was calculated as the % of prescribed treatment actually completed: total hours of game play since baseline divided by the total prescribed hours (based on intended dose of 1 hour a day, 7 days per week) since baseline.
Time Frame: Entire study period, up to 16 weeks
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: % of prescribed treatment completed
Arm/Group | Binocular Treatment Younger | Binocular Treatment Older Cohort
Number analyzed (Participants) | 176 | 38
% of prescribed treatment completed | 46 [20 to 72] | 21 [13 to 38]

19. Other Pre Specified Outcome: Percentage of Participants Reporting >75% of Prescribed Treatment Completed (Subjective Measures of Adherence)
Description: Participants who were randomly assigned to binocular treatment were prescribed 1 hour of game play per day, 7 days a week while those assigned to the patching group were prescribed 2 hours of daily patching, 7 days per week.
  Parents were asked to record the amount of time that the participant played the binocular game (binocular treatment group) or wore the patch (patching group) each day on a calendar.
  At each study visit, the investigator estimated the frequency and duration of treatment that the participant completed based on the parent-reported calendars and discussion with the participant and/or parent(s). For analysis, the percentage of prescribed treatment completed was calculated as the total number of reported hours of treatment completed since baseline divided by the total number of prescribed hours (refer to the intended treatment dose/frequency listed above) since baseline.
Time Frame: 16 Weeks from baseline
Population: The descriptive analysis included data from participants who completed the 16-week visit within the predefined analysis window (14 to <20 weeks after randomization).
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger | Binocular Treatment Older Cohort | Patching Treatment Older Cohort
Number analyzed (Participants) | 177 | 186 | 39 | 56
Participants | 118 | 172 | 24 | 42

20. Other Pre Specified Outcome: Participants Who Received Non-protocol, Alternative Treatment During the Study
Description: Participants who were randomly assigned to binocular treatment were prescribed 1 hour of game play per day, 7 days a week while those assigned to the patching group were prescribed 2 hours of daily patching, 7 days per week.
  The number of participants who received non-protocol, alternative treatment was tabulated by treatment group.
Time Frame: Entire study period, up to 16 weeks
Population: All randomized participants in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger | Binocular Treatment Older Cohort | Patching Treatment Older Cohort
Number analyzed (Participants) | 190 | 195 | 40 | 60
Participants | 4 | 0 | 0 | 0

21. Other Pre Specified Outcome: Safety Analysis: Distribution of the Change in Fellow-eye Visual Acuity From Baseline
Description: Monocular distance visual acuity (VA) in current refractive correction (if required) in each eye by a certified examiner using the electronic ATS-HOTV visual acuity protocol for children <7 years and the E-ETDRS visual acuity protocol for children ≥ 7 years on a study-certified acuity tester displaying single surrounded optotypes. The change in visual acuity is analyzed as logMAR lines for the younger cohort and as letters for the older cohort.
Time Frame: 16-week visit
Population: Participants who completed the 16-week visit (regardless of whether or not the visit was completed within the pre-specified analysis window).
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger | Binocular Treatment Older Cohort | Patching Treatment Older Cohort
Number analyzed (Participants) | 182 | 188 | 39 | 58
Participants
  2 lines (10-14 letters) better | 6 | 2 | 0 | 2
  1 line (5-9 letters) better | 36 | 30 | 10 | 9
  0 line (within 4 letters) | 128 | 133 | 29 | 46
  1 line (5-9 letters) worse | 11 | 22 | 0 | 1
  2 lines (10-14 letters) worse | 1 | 1 | 0 | 0

22. Other Pre Specified Outcome: Safety Analysis: Change in Fellow-eye Visual Acuity From Baseline (Younger Cohort)
Description: Monocular distance visual acuity (VA) in current refractive correction (if required) in each eye by a certified examiner using the electronic Amblyopia Treatment Study single-surround HOTV (ATS-HOTV) visual acuity protocol for children <7 years and the Electronic Early Treatment Diabetic Retinoscopy Study (E-ETDRS) visual acuity protocol for children ≥ 7 years on a study-certified acuity tester displaying single surrounded optotypes.
  For the younger cohort, the level of visual acuity is analyzed in the log of the Minimum Angle of Resolution (logMAR) scale (approximate range: -0.2 to 1.7) such that higher scores indicate poorer VA. Change in VA is computed as logMAR lines (positive values indicate improvement), defined as the difference between the enrollment and 16-week acuities (logMAR) multiplied by 10.
  For this safety analysis, the change in fellow-eye visual acuity (logMAR lines) was computed by treatment group, adjusting for baseline visual acuity.
Time Frame: 16-week visit
Population: as for outcome 21
Measure: Mean (95% Confidence Interval); unit: logMAR lines
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger
Number analyzed (Participants) | 182 | 188
logMAR lines | 0.30 [0.20 to 0.40] | 0.14 [0.04 to 0.24]
Statistical Analysis 1: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; The treatment group difference in the change in fellow-eye visual acuity from baseline to 16 weeks (logMAR lines) was evaluated in an analysis of covariance model, adjusted for baseline fellow-eye visual acuity; Test type: Superiority; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [0.02 to 0.30] — A 95% confidence interval was computed on the adjusted treatment group difference (binocular treatment - patching) in mean change in fellow-eye visual acuity from baseline to 16 weeks. Positive values favor the binocular treatment group

23. Other Pre Specified Outcome: Safety Analysis: Change in Fellow-eye Visual Acuity From Baseline (Older Cohort)
Description: Monocular distance visual acuity (VA) in current refractive correction (if required) in each eye by a certified examiner using the Electronic Early Treatment Diabetic Retinoscopy Study (E-ETDRS) visual acuity protocol for children ≥ 7 years on a study-certified acuity tester displaying single surrounded optotypes.
  For the analyses in the older cohort, the level of VA is measured as letter scores (approximate range: 0 to 97 letters, lower scores indicate poorer VA) and change in VA from baseline is measured in letters (positive values indicate improvement), defined as the difference in letter scores between enrollment and follow-up.
  The change in fellow-eye visual acuity (letters) from baseline (positive values indicate improvement) was computed by treatment group, adjusting for baseline visual acuity.
Time Frame: 16-week visit
Population: as for outcome 21
Measure: Mean (95% Confidence Interval); unit: Letters
Arm/Group | Binocular Treatment Older Cohort | Patching Treatment Older Cohort
Number analyzed (Participants) | 39 | 58
Letters | 2.2 [1.2 to 3.1] | 2.0 [1.3 to 2.8]
Statistical Analysis 1: Comparison: Binocular Treatment Older Cohort vs Patching Treatment Older Cohort; An analysis of covariance (ANCOVA) model was used to compute the treatment group difference in the mean change in fellow-eye visual acuity (letters) from baseline to 16 weeks, adjusting for baseline visual acuity. A 2-sided 95% confidence interval was computed on the adjusted treatment group difference; Test type: Superiority; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-1.1 to 1.3] — A 95% confidence interval was computed on the treatment group difference (binocular treatment - patching) of the adjusted mean change in fellow-eye visual acuity from baseline to 16 weeks

24. Other Pre Specified Outcome: Safety Analysis: Development of a New Tropia and/or Worsening of a Pre-existing Deviation by 10 pd
Description: Ocular alignment will be assessed in current refractive correction by the cover/uncover test, simultaneous prism and cover test (SPCT), and prism and alternate cover test (PACT) in primary gaze at distance (3 meters) and at near (1/3 meter).
  Participants were classified according to whether they met the any of the following criteria at the 16-week visit: development of a new tropia (measured by SPCT) and/or worsening of a pre-existing deviation by 10 prism diopters (pd) measured by SPCT.
Time Frame: 16 weeks
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger | Binocular Treatment Older Cohort | Patching Treatment Older Cohort
Number analyzed (Participants) | 182 | 188 | 39 | 58
Participants | 16 | 11 | 3 | 3
Statistical Analysis 1: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; Fisher's exact test was used to perform the treatment group comparison of the proportion of participants who developed a new ocular deviation and/or worsening of a pre-existing ocular deviation by 10 prism diopters at the 16-week visit; Test type: Superiority; p = 0.32, Fisher Exact
Statistical Analysis 2: Comparison: Binocular Treatment Older Cohort vs Patching Treatment Older Cohort; [analysis description as in outcome 24, analysis 1]; Test type: Superiority; p = 0.68, Fisher Exact

25. Other Pre Specified Outcome: Safety Analysis: Distribution of Diplopia Frequency at 16 Weeks (Parent-reported)
Description: A standardized questionnaire was administered to participants and their parents to assess the presence and frequency of any diplopia since the last study visit.
Time Frame: 16 weeks
Population: Participants whose parent completed a 16-week diplopia assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger | Binocular Treatment Older Cohort | Patching Treatment Older Cohort
Number analyzed (Participants) | 182 | 187 | 38 | 57
Participants
  No diplopia | 176 | 185 | 37 | 56
  Diplopia: Less than once a week | 5 | 0 | 1 | 1
  Diplopia: Once a week | 1 | 2 | 0 | 0
  Diplopia: Once a day | 0 | 0 | 0 | 0
  Diplopia: Up to 10 times a day | 0 | 0 | 0 | 0
  Diplopia: >10 times a day | 0 | 0 | 0 | 0
  All the time | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; The Fisher exact test was used to compare the percentage of parents who reported that their child had experienced diplopia (yes/no) at the 16-week visit by treatment group; Test type: Superiority; p = 0.17, Fisher Exact
Statistical Analysis 2: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; The frequency of diplopia, across categories of diplopia, was compared between the treatment groups using the Cochran-Armitage trend test; Test type: Superiority; p = 0.48, Cochran-Armitage trend test
Statistical Analysis 3: Comparison: Binocular Treatment Older Cohort vs Patching Treatment Older Cohort; [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p > 0.99, Fisher Exact
Statistical Analysis 4: Comparison: Binocular Treatment Older Cohort vs Patching Treatment Older Cohort; [analysis description as in outcome 25, analysis 2]; Test type: Superiority; p > 0.99, Cochran-Armitage trend test

26. Other Pre Specified Outcome: Safety Analysis: Distribution of Diplopia Frequency at 16 Weeks (Participant-reported)
Description: as for outcome 25
Time Frame: 16 weeks
Population: Participants who completed a 16-week diplopia assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger | Binocular Treatment Older Cohort | Patching Treatment Older Cohort
Number analyzed (Participants) | 182 | 188 | 39 | 58
Participants
  No diplopia | 166 | 181 | 37 | 56
  Diplopia: Less than once a week | 5 | 3 | 0 | 0
  Diplopia: Once a week | 5 | 3 | 2 | 1
  Diplopia: Once a day | 2 | 1 | 0 | 0
  Diplopia: Up to 10 times a day | 3 | 0 | 0 | 1
  Diplopia: >10 times a day | 0 | 0 | 0 | 0
  All the time | 1 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; The Fisher exact test was used to compare the percentage of participants who reported diplopia (yes/no) at the 16-week visit by treatment group; Test type: Superiority; p = 0.05, Fisher Exact
Statistical Analysis 2: Comparison: Binocular Treatment Younger vs Patching Treatment Younger; [analysis description as in outcome 25, analysis 2]; Test type: Superiority; p = 0.02, Cochran-Armitage trend test
Statistical Analysis 3: Comparison: Binocular Treatment Older Cohort vs Patching Treatment Older Cohort; [analysis description as in outcome 26, analysis 1]; Test type: Superiority; p > 0.99, Fisher Exact
Statistical Analysis 4: Comparison: Binocular Treatment Older Cohort vs Patching Treatment Older Cohort; [analysis description as in outcome 25, analysis 2]; Test type: Superiority; p > 0.99, Cochran-Armitage trend test

27. Other Pre Specified Outcome: Safety Analysis: Distribution of Maximum Frequency of Diplopia Reported Across Follow-up (Parent-reported)
Description: as for outcome 25
Time Frame: Across study follow-up visits, up to 16 weeks
Population: Participants whose parent completed a diplopia assessment at any follow-up visit (4-week, 8-week, 12-week, 16-week)
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger | Binocular Treatment Older Cohort | Patching Treatment Older Cohort
Number analyzed (Participants) | 182 | 188 | 39 | 58
Participants
  No diplopia | 172 | 182 | 38 | 54
  Diplopia: Less than once a week | 6 | 4 | 0 | 2
  Diplopia: Once a week | 2 | 1 | 1 | 1
  Diplopia: Once a day | 2 | 0 | 0 | 1
  Diplopia: Up to 10 times a day | 0 | 1 | 0 | 0
  Diplopia: >10 times a day | 0 | 0 | 0 | 0
  All the time | 0 | 0 | 0 | 0

28. Other Pre Specified Outcome: Safety Analysis: Distribution of Maximum Frequency of Diplopia Reported Across Study Follow-up (Participant-reported)
Description: as for outcome 25
Time Frame: Across study follow-up visits, up to 16 weeks
Population: Participants who completed a diplopia assessment at any follow-up visit (4-week, 8-week, 12-week, 16-week) during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger | Binocular Treatment Older Cohort | Patching Treatment Older Cohort
Number analyzed (Participants) | 182 | 188 | 39 | 58
Participants
  No diplopia | 153 | 167 | 36 | 50
  Diplopia: Less than once a week | 6 | 10 | 1 | 1
  Diplopia: Once a week | 10 | 4 | 0 | 3
  Diplopia: Once a day | 8 | 5 | 2 | 3
  Diplopia: Up to 10 times a day | 3 | 2 | 0 | 1
  Diplopia: >10 times a day | 1 | 0 | 0 | 0
  All the time | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Binocular Treatment Younger | Patching Treatment Younger | Binocular Treatment Older | Patching Treatment Older
Serious Adverse Events (participants affected / at risk) | 0/190 | 0/195 | 0/40 | 0/60
Other Adverse Events (participants affected / at risk) | 0/190 | 0/195 | 0/40 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No